CLINICAL TRIAL: NCT00435084
Title: An Open Phase I/II Clinical Study Assessing the Safety and Tolerability of APO866 in Patients With Refractory B-cell Lymphocytic Leukaemia Not Amenable to Allogeneic Hemopoietic Stem Cell Transplantation
Brief Title: A Phase I/II Study to Assess the Safety and Tolerability of APO866 for the Treatment of Refractory B-CLL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP3005; EudraCT number 2006-002850-31
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2013-11

CONDITIONS: B-cell Chronic Lymphocytic Leukemia
Keywords: Refractory B-CLL; phase I/II; CD38
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — N-(4-(1-benzoylpiperidin-4-yl)butyl)-3-(pyridin-3-yl)acrylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm mono therapy (Experimental): APO866 will be administered by civ infusion at 0.126 mg/m2/hr for 4 consecutive days (96 hours). This constitutes 1 cycle.
  Interventions: Drug: APO866

INTERVENTIONS:
Drug: APO866

SUMMARY:
This phase I/II study is designed to determine the safety and tolerability of APO866 for the treatment of refractory B-CLL not amenable to aHSCT. APO866 has shown to induce growth inhibition in cultures of a wide variety of human hematological malignant cells as well as in models with subcutaneously implanted human tumors. APO866 was considered to be safe and well-tolerated in a phase I study that treated 24 patients with advanced cancer. APO866 is administered by intravenous infusion continuously for 96 hours and is repeated every 4 weeks. In this study patients will receive only one cycle of treatment and the study endpoints will be evaluated 4 weeks after the start of infusion. Patients will be followed up for 12 weeks for safety.

DETAILED DESCRIPTION:
B-CLL is one of the most common types of leukemia, remains incurable, and has only limited therapeutic options available including alkylating agents and fludarabine. The identification of new, selective, and non-toxic forms of therapy for patients with B-CLL is therefore a high priority.

APO866 is a novel drug that induces cell death by specifically inhibiting the biosynthesis of NAD+ from niacinamide, which is essential for the cellular metabolism, protein modification and messenger synthesis. APO866 is not subject to the commonly known mechanisms of MDR. Its activity is cell cycle independent. APO866 exerted high anti-tumor activity on a broad range of different tumor cells derived from both human solid cancers and leukemias in vitro, including CD38- and CD38+ cell lines, and on a large number of human xenografts in nude mice and rats in vivo. Hematologic cancer cells were highly sensitive to APO866 (lower than 6 nM). Lymphocytes are the most sensitive normal cells to APO866 resulting in lymphocytopenia and reticulocytopenia in rats and monkeys. Furthermore, APO866 may have anti-angiogenic properties as shown in vivo and dose-dependent decrease of VEGF levels in patients treated in the phase I study.

It is unclear why CD38 positivity is associated with a short patient survival and poor responsiveness to chemotherapy. It is possible that CD38 expression confers to B-CLL of a more malignant cellular phenotype. This seems plausible given that the antigen has an important role as a modulator of intracellular signaling and that cross-linking of CD38 up-regulates BCL-2 and inhibits apoptosis in normal mature B cells. Indeed, CD38/CD3l interactions lead to increased B-CLL proliferation and survival. This study has been designed to recruit patients with progressive or refractory B-CLL of whom, in line with the literature, about 50% will be CD38+.

We hypothesize that CD38+ lymphocytes will be more sensitive to the APO866 therapy due to increased intracellular NAD+ consumption as substrate for the PARP dependent DNA repair (instable genome, proliferation). However, CD38+ and CD38- B-CLL cells seem to be equally sensitive to APO866 in vitro. In addition, decreased intracellular NAD+ levels will reduce the anabolism of cADPR. CD38+ can catalyze the synthesis of cADPR from NAD+ and can further hydrolyze cADPR to ADP-ribose.85,86,87 The cADPR is a potent Ca++-mobilizing activator and a potential endogenous regulator.88 The ability of cADPR to release Ca++ from intracellular pools is thought to be part of CD38-mediated signalling pathways that result in cell growth, apoptosis, and differentiation.

APO866 was investigated in 24 patients with advanced cancers in a phase I study aiming to determine the DLT and MTD. Treatment was well tolerated and safe. The unique DLT was thrombocytopenia. At dose levels higher than 0.036 mg/m2/hr CTC grade III lymphocytopenia, not thought to be clinically relevant, preceded all other toxicities. The recommended dose for phase II studies of APO866 is 0.126 mg/m2/hr administered by civ infusion for 4 consecutive days every 4 weeks. This dose was selected because of its safety profile, and the translational observation that Css of APO866 at MTD was similar or higher as compared to the concentrations at which efficacy was established in vitro and in vivo. In addition, a transient decrease of serum VEGF levels, a surrogate marker of angiogenesis, was observed within 96 hrs after the start of treatment in 9 out of 11 patients treated at MTD and the 0.144 mg/m2/hr dose level of APO866

This forms the rationale to conduct a "Proof of concept" study of APO866, administered at the recommended dose in patients with progressive refractory B-CLL non-eligible for aHSCT, either CD38- or CD38+.

ELIGIBILITY:
Inclusion Criteria:

* Immunophenotypic (monoclonal population of mature CD5+, CD19+, CD23+) confirmed diagnosis of B-CLL
* Diagnosis of progressive symptomatic B-CLL requiring therapy (Revised NCI-sponsored Working Group guidelines for CLL
* Relapsed or refractory disease or intolerant to ≥ 2 prior systemic therapy. (containing either a purine analog or an alkylating agent). Patient is not amenable to aHSCT
* ECOG Performance Status < 2
* Age > 18 years, of either sex
* Female patients with childbearing potential must be using a hormonal contraceptive, intra uterine device, diaphragm with spermicide or condom with spermicide for the duration of the study. Women of childbearing potential must have a negative serum or urinary hCG pregnancy test within 7 days prior to Study Day 1 (SD1)
* Male patients, who are not surgically sterile, must use a condom with spermicide for the duration of the study and 3 months thereafter
* Have given written informed consent, prior to any study related procedure not part of the patient's normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

* Have participated in any other investigational study or received an experimental therapeutic procedure considered to interfere with the study in the 4 weeks preceding SD1
* Use of prohibited medication due to CYP3A4 metabolism of APO866, as specified in Section 6.6.2. concomitant use of these drugs will not be allowed during the study
* Uncontrolled medical conditions, requiring surgical or pharmacological treatment (exceptions must be approved by the Medical Responsible of the study)
* Active infection requiring systemic antibiotics
* Serious concomitant disease (e.g. significant cardiac disease)
* History of second cancer that was treated with curative intent and in complete remission for < 5 years, with the exception of basal cell carcinoma or cervical cancer in situ
* Inadequate bone marrow function: platelets < 75x10^9/L without transfusion in the preceding 2 weeks, ANC < 1,0x10^9/L without growth factor support, abnormal coagulation APTT and PT
* Platelet-refractory state due to platelet alloimmunization
* Inadequate liver function: total bilirubin > 1.5x upper limit of normal values (ULN), AST, ALT, or alkaline phosphatase > 2.5x ULN
* Inadequate renal function: serum creatinine > 1.5x ULN
* Retinopathy, history of retinal laser surgery, or an ERG < 50% of normal
* Pregnant or lactating female
* Known allergy to reagents in the study drug (APO866 or propylene glycol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of APO866 in patients with refractory B-CLL not amenable to allogeneic HSCT | 1 month

SECONDARY OUTCOMES:
To determine the effect on the number of circulating leukemic after treatment as compared to baseline | 1 month
To determine the effect on the number of CD38+ after treatment as compared to baseline | 1 month
Correlative analysis on in vivo and in vitro sensitivity of leukemic cells, CD38 expression of leukemic cells and clinical outcome, immunophenotype and clinical outcome | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hillmen, MD PhD, Principal Investigator — Department of Heamatology, D Floor, Brotherton Wing, Leeds General Infirmary, Great George street, Leeds LS1 3EX; René Goedkoop, MD, Study Director — Apoxis SA, 18-20 Avenue de Sévelin, 1004 Lausanne, Switzerland
Locations (4):
- United Kingdom (4):
  - Department of Heamtology, Cardiff and Vale NHS Trust, Cardiff
  - Department of Heamtology, Leeds General Infirmary, Leeds
  - Department of Heamtology, Bart's and the London NHS Trust, London
  - Department of Heamtology, University Hospital of NHS Trust, Nottingham